CLINICAL TRIAL: NCT00194857
Title: A Randomized Clinical Trial Comparing Two Management Strategies for Treatment of Neutropenia and Anemia Associated With Pegylated Interferon Plus Ribavirin Treatment of Compensated Chronic Hepatitis C in Adult Subjects Infected With HIV.
Brief Title: Treatment of Anemia and Neutropenia in HIV/HCV Coinfected Patients Treated With Pegylated Interferon and Ribavirin
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Schering-Plough (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03850-001; 0801-858
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Anemia; Neutropenia; Hepatitis C Virus; HIV Infections
Keywords: anemia; dose reduction; neutropenia; hepatitis C virus; human immunodeficiency virus
MeSH Terms: conditions — Anemia; Neutropenia; Hepatitis C; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Erythropoietin

INTERVENTIONS:
Drug: erythropoietin, GCSF

SUMMARY:
This study is designed to test two separate strategies for treatment of anemia (low hemoglobin) and neutropenia (low white blood cells) in HIV/HCV coinfected patients who are being treated with pegylated interferon and ribavirin.

DETAILED DESCRIPTION:
This is a multi-center, randomized, open-labeled trial in subjects co-infected with hepatitis C (HCV) and human immunodeficiency virus type 1 (HIV-1) who are naïve to anti-HCV therapy. Subjects will receive PEG interferon alfa-2b (PEG-IFN) 1.5 mcg/kg/week administered once weekly plus ribavirin (RBV) 13 + 2 mg/kg/day. The goal of this study is to evaluate two different treatment options for anemia and neutropenia associated with the initiation of pegylated interferon and ribavirin. This will result in completion of therapy, and possibly a better viral sustained response.

ELIGIBILITY:
Inclusion Criteria:

* hemoglobin > 11
* absolute neutrophil count >1,200
* naive to peg interferon and ribavirin

Exclusion Criteria:

* Prior treatment for hepatitis C
* Pregnant or nursing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
change in hemoglobin
change in absolute neutrophil count

SECONDARY OUTCOMES:
HCV RNA
depression
fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Talal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Derived] Talal AH, Liu RC, Zeremski M, Dimova R, Dove L, Pearce D, Hassanein T, Doonquah L, Aboulafia D, Rodriguez J, Bonilla H, Galpin J, Aberg JA, Johnston B, Glesby MJ, Jacobson IM. Randomized trial comparing dose reduction and growth factor supplementation for management of hematological side effects in HIV/hepatitis C virus patients receiving pegylated-interferon and ribavirin. J Acquir Immune Defic Syndr. 2011 Nov 1;58(3):261-8. doi: 10.1097/QAI.0b013e3182324af9. PMID 21876446